CLINICAL TRIAL: NCT06243952
Title: Brain Controlled Spinal Cord Stimulation In Participants With Spinal Cord Injury For Lower Limb Rehabilitation
Acronym: Think2Go
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Prof., Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Think2Go
Record Dates: First submitted 2023-12-11; First posted 2024-02-06 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Paraplegia
Keywords: Spinal cord stimulation; Brain computer interface; Brain spine interface
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Intervention Model Description: monocentric, single-arm, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): All participants receive the same intervention.
  Interventions: Device: ARC-BSI Lumbar system

INTERVENTIONS:
Device: ARC-BSI Lumbar system — Implantation of a 64 channel - ECoG array over the sensory motor cortex of the lower limbs, combined with an implantation of 16 channel spinal cord stimulation system over the lumbar region. The decoded motor intentions are driving the implanted spinal cord stimulation system. Brain-controlled spinal cord stimulation is used for training and rehabilitation to recover voluntary movements.

SUMMARY:
The purpose of this clinical study is to evaluate the preliminary safety and effectiveness of using a cortical recording device (ECoG) combined with lumbar targeted epidural electrical stimulation (EES) of the spinal cord to restore voluntary motor functions of lower limbs in participants with chronic spinal cord injury suffering from mobility impairment.

The goal is to establish a direct bridge between the motor intention of the participant and the the spinal cord below the lesion, which should not only improve or restore voluntary control of legs movement and support immediate locomotion, but also promote neurological recovery when combined with neurorehabilitation.

DETAILED DESCRIPTION:
In a current first-in-human clinical trial, called STIMO (ClinicalTrials.gov, NCT02936453), Electrical Epidural Stimulation (EES) of the spinal cord is applied to enable individuals with chronic severe spinal cord injury (SCI) to complete intensive locomotor neurorehabilitation training. In this clinical feasibility study, EES immediately enhances walking function and, with repeated use as part of the EES-assisted neurorehabilitation program, improves leg motor control and neurological recovery in severe SCI participants to a certain extent. Linking brain activity to spinal stimulation, as shown in preclinical and clinical studies, enhances usability of EES and neurological recovery.

Clinatec (CEA, Grenoble, France) has developed an implantable electrocorticogram (ECoG) recording device with a 64-channel epidural electrode array called WIMAGINE capable of recording electrical signals from the motor cortex for an extended period and with a high signal to noise ratio. This ECoG-based system allowed tetraplegic patients to control an exoskeleton (Clinicaltrials.gov, NCT 02550522) with up to 8 degrees of freedom for the upper limb control. This device has been implanted in 5 chronic participants so far; one of them has been using this system both at the hospital and at home for more than 3 years.

The ECoG WIMAGINE technology has been combined with EES in the current first-in-human clinical trial STIMO-BSI (Brain Spine Interface) (Clinicaltrials.gov, NTC04632290): with the WIMAGINE technology, cortical motor intentions for leg movements are recorded, and real-time decoding translates brain signals into EES commands. This digital bridge empowered a chronic SCI participant, who has been part of the STIMO clinical trial, to regain leg motor control by volitional fine-tuned EES amplitudes enabling standing, walking and adapting to diverse terrains, demonstrating the efficacy of the BSI. Moreover, BSI-assisted neurorehabilitation mediated neurological improvements after three years of stable performance of the patient, that persisted even when the BSI was switched off.

In this study, the investigators will assess the preliminary safety and effectiveness of ECoG-controlled EES in individuals with chronic SCI who have not previously participated in STIMO clinical trial, to establish a direct bridge between the motor intention and the spinal cord below the lesion. This could improve or restore voluntary control of legs movement as well as promote neurological recovery when combined with neurorehabilitation. The WIMAGINE ECoG system will be coupled with the ARC-IM purpose-built spinal cord stimulation technology in the ARC-BSI Lumbar system. An equivalent technology (ARC-BSI Cervical system) is currently used in the ongoing UP2 clinical study (Clinicaltrials.gov, NCT05665998) for upper limb rehabilitation in patients with cervical spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide Informed Consent as documented by signature (Appendix Informed Consent Form) prior to any study-related procedures,
2. Must be at least 18 years old and no older than 60 years old at the time of enrolment,
3. Must be suffering from non-progressive traumatic spinal cord injury,
4. Must be graded A, B, C, or D in the American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification,
5. Must have completed primary standard of care rehabilitation,
6. Must have stable medical, physical and psychological condition as considered by the investigator,
7. Must be lesioned at T10 or above, based on AIS level determination by the investigator, with preservation of conus function,
8. Must have sustained the injury at least 12 months before signing the consent form,
9. Must have residual upper limb function (capable of using a manual wheelchair),
10. Must be able to understand and interact with the study team in French or English,
11. Must agree to comply in good faith with all conditions of the study and to attend all scheduled appointments,
12. Must use safe contraception for women of childbearing capacity.

Exclusion Criteria:

1. Must not be pregnant nor breast feeding,
2. Must not have the intention to become pregnant during the course of the study,
3. Must not have brain damage,
4. Must not have history of epilepsy,
5. Must not have participated in another clinical study using drugs or medical devices within the 30 days preceding and during the present study,
6. Must not have previously been injected with stem cells in the spinal cord,
7. Must not have any hematological disorders with increased risk for surgical intervention,
8. Must not require ventilator support,
9. Must not have limitation of walking function based on accompanying (Central Nervous System (CNS)) disorders (systemic malignant disorders, cardiovascular disorders restricting physical training, peripheral nerve disorders),
10. Must not suffer from spinal cord injury from other etiology than traumatic (ischemic, tumoral, autoimmune, etc.),
11. Must not display spinal stenosis or post traumatic damage at location of implantation,
12. Must not require the use of an intrathecal baclofen pump,
13. Must not be implanted with a device such as pacemakers or defibrillators,
14. Must not have any indication that would require Magnetic Resonance Imaging (MRI),
15. Must not suffer from congenital nor acquired lower limb abnormalities (affection of joints or bones).
16. Must not be the investigator himself, his/her family members, employees or other dependent persons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Preliminary safety | Through study completion (implantation up to end of study - average of 1 year)
  Occurrence of Serious Adverse Events (SAE) and Adverse Events (AE) that are deemed related or possibly related to the procedure or to the ARC-BSI Lumbar System.

SECONDARY OUTCOMES:
10 Meters Walk Test (10MWT) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Clinical measure to assess walking speed (in m/s) over 10 meters.
6 Minutes Walk Test (6MWT) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Submaximal test to assess endurance during 6 minutes of walking.
Timed Up and Go (TUG) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Timed test of functional mobility (stand-up, walk, turn around, sit-down)
Walking Index for Spinal Cord Injury (WISCI II) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Clinical tool to capture the extent and nature of assistance a person with SCI requires to walk, on an ordinal scale of 20 levels, from the most severe impairment (level 0) to the least severe impairment (level 20).
Berg Balance Scale (BBS) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Test to measure static balance and fall risk among adults by assessing the performance at functional tasks with a 14-item scale. From 0 to 56, higher scores mean a better outcome.
Neuromuscular Recovery Scale (NRS) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Clinical assessment tool that quantifies recovery from spinal cord injury by measuring functionally relevant motor tasks without compensation strategies. The trunk and lower extremities recovery will be assessed on 10 items.
Spinal Cord Injury Functional Ambulation Inventory (SCI-FAI) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Observational gait assessment that includes 3 key domains of walking function, where 0 is the minimum and worst outcome: gait parameters (maximum score of 20 points), assistive devices (each limb scored individually - maximum score of 14 points), temporal distance (maximum score of 5 points).
EMG-based Gait Analysis | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Evaluation of locomotion parameters during different walking tasks (walking on a treadmill, walking over ground, "parcours" with obstacles and different surfaces), assessing biomechanics of movement through the acquisition of electromyographic data (electrical activity, in millivolts, associated to muscular fibers contraction) with placement of wearable sensors on the legs muscles.
Kinematics-based Gait Analysis | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Evaluation of locomotion parameters during different walking tasks (walking on a treadmill, walking over ground, "parcours" with obstacles and different surfaces), assessing biomechanics of movement through the acquisition of kinematic data (displacement in the 3 directions of space, in millimeters) with placement of wearable markers on the legs joints.
Presence of visible movements during single joints movements attempts, measured in angular displacement of the joint (degrees, °) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Assessment of the presence of visible movements for right and left hip (flexion), ankle (dorsiflexion) and knee (extension).
Spasticity assessment (Modified Ashworth Scale - MAS) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Resistance of a muscle to a passive range of motion about a single joint (6-points nominal scale).
ASIA impairment scale - International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Clinical examination used to assess the motor and sensory impairment and severity of a spinal cord injury.
Somato-Sensory Evoked Potential (SSEP) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Electrophysiological measure that evaluates the transmission of electrical pulses resulting from electrical stimulation of the dorsal roots of the spinal cord through the ARC-IM stimulation lead, by recording the cortical response with the WIMAGINE implant.

OTHER OUTCOMES:
WHOQOL-BREF (World Health Organization Quality of Life) | Pre-implantation (up to 4 weeks before implantation), during BSI configuration (at 4 weeks and and lasting up to 2 weeks), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Quality of life assessment. From 0 to 100, higher scores mean a better outcome.
PIADS (Psychosocial Impact of Assistive Device Scale) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  26-item, self-report questionnaire to assess the effects of an assistive device on functional independence. Each item is scored from -3 (decreases) to 3 (increases).
SCIM III (Spinal Cord Independence Measure) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  19-items-measure of the functional independence of individuals with spinal cord injury, organized in 3 subscales: self-care, respiration and sphincter management, and mobility.
GAS (Goal Attainment Scaling) | Pre-implantation (up to 4 weeks before implantation), post-rehabilitation (at 24 weeks and lasting up to 2 weeks) and post-remote follow up (at 1 year and lasting up to 2 weeks).
  Method of scoring the extent to which patients individual goals are achieved in the course of intervention. Six patient-therapist goal will be defined before treatment and a measurable scale for each goal will be set up, specifying, for each patient, a transformation of his overall goal attainment into a standardized T-score.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Bonizzato M, Pidpruzhnykova G, DiGiovanna J, Shkorbatova P, Pavlova N, Micera S, Courtine G. Brain-controlled modulation of spinal circuits improves recovery from spinal cord injury. Nat Commun. 2018 Aug 1;9(1):3015. doi: 10.1038/s41467-018-05282-6. PMID 30068906
- [Background] Capogrosso M, Wenger N, Raspopovic S, Musienko P, Beauparlant J, Bassi Luciani L, Courtine G, Micera S. A computational model for epidural electrical stimulation of spinal sensorimotor circuits. J Neurosci. 2013 Dec 4;33(49):19326-40. doi: 10.1523/JNEUROSCI.1688-13.2013. PMID 24305828
- [Background] Lorach H, Galvez A, Spagnolo V, Martel F, Karakas S, Intering N, Vat M, Faivre O, Harte C, Komi S, Ravier J, Collin T, Coquoz L, Sakr I, Baaklini E, Hernandez-Charpak SD, Dumont G, Buschman R, Buse N, Denison T, van Nes I, Asboth L, Watrin A, Struber L, Sauter-Starace F, Langar L, Auboiroux V, Carda S, Chabardes S, Aksenova T, Demesmaeker R, Charvet G, Bloch J, Courtine G. Walking naturally after spinal cord injury using a brain-spine interface. Nature. 2023 Jun;618(7963):126-133. doi: 10.1038/s41586-023-06094-5. Epub 2023 May 24. PMID 37225984
- [Background] Benabid AL, Costecalde T, Eliseyev A, Charvet G, Verney A, Karakas S, Foerster M, Lambert A, Moriniere B, Abroug N, Schaeffer MC, Moly A, Sauter-Starace F, Ratel D, Moro C, Torres-Martinez N, Langar L, Oddoux M, Polosan M, Pezzani S, Auboiroux V, Aksenova T, Mestais C, Chabardes S. An exoskeleton controlled by an epidural wireless brain-machine interface in a tetraplegic patient: a proof-of-concept demonstration. Lancet Neurol. 2019 Dec;18(12):1112-1122. doi: 10.1016/S1474-4422(19)30321-7. Epub 2019 Oct 3. PMID 31587955